CLINICAL TRIAL: NCT04954729
Title: Association of Processing Speed Dysfunction and Brain Functional Abnormality in Childhood Epilepsy With Centrotemporal Spikes
Brief Title: Association of Processing Speed Dysfunction and Brain Functional Abnormality in ECTS
Status: Completed | Type: Observational
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Other Study IDs: 2019-266
Record Dates: First submitted 2021-07-06; First posted 2021-07-08 (Actual); Last update posted 2021-07-08 (Actual); Status verified 2021-07

CONDITIONS: Epilepsy, Rolandic
Keywords: Processing speed; Epilepsy; Positron emission tomography; Functional magnetic resonance imaging
MeSH Terms: conditions — Epilepsy, Rolandic; Epilepsy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Experimental Group: The experimental group underwent neuropsychological testing, 18F-FDG PET/CT, 3T resting state fMRI examinations.
- MRI Control Group: The MRI control group underwent neuropsychological testing and 3T resting state fMRI examinations
- PET Control Group: The PET control group underwent 18F-FDG PET/CT examination

SUMMARY:
Epilepsy with centrotemporal spikes (ECTS) is the most common epilepsy syndrome in children. Language impairment has been widely investigated in patients with ECTS, but little is known about the cognitive dysfunction of processing speed and its neuroimaging mechanism.

DETAILED DESCRIPTION:
OBJECTIVE To investigate the processing speed dysfunction in patients with ECTS, and the associated brain functional abnormality using functional magnetic resonance imaging (fMRI) and 18F-fluorodeoxyglucose (18F-FDG) positron emission tomography (PET).

DESIGN, SETTING, AND PARTICIPANTS This study prospectively enrolled ECTS patients (n = 28) from June 2019 and June 2021. Twenty age- and gender- matched healthy children and another twenty children with extracranial tumors were enrolled as controls. Patients with ECTS and healthy controls underwent neuropsychological testing and fMRI examination. In addition, ECTS patients and children with extracranial tumors underwent 18F-FDG PET examination.

ELIGIBILITY:
Inclusion Criteria:

* (a) age between 6 and 18 years; (b) 18F-FDG PET examination more than 48 h since the last seizure, (c) no structural abnormalities associated with epilepsy detected on routine MRI

Exclusion Criteria:

* (a) any history of other neurological or psychiatric disorders; (b) pre-scan plasma glucose level > 120 mg/dl before 18F-FDG PET/CT examination;(c) any contraindications for MRI examination ; (d) head movement (translation > 3 mm or rotation > 3 degree ) during MRI examination

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Pediatric patients with childhood epilepsy with centrotemporal spikes
Sampling Method: Non-Probability Sample
Enrollment: 68 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2021-06-01 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Processing speed index | Through study completion, about 2 years
  Processing speed index was measured according to Wechsler Intelligence Scale for Children
Standardized uptake value ratio | Through study completion, about 2 years
  Standardized uptake value ratio was measured from 18F-FDG PET for brain glucose metabolism
Functional connectivity | Through study completion, about 2 years
  Functional connectivity was measured from fMRI for brain regional interactions

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Nuclear Medicine and PET/CT Center, The Second Affiliated Hospital, School of Medicine, Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Li Y, Zhang T, Feng J, Qian S, Wu S, Zhou R, Wang J, Sa G, Wang X, Li L, Chen F, Yang H, Zhang H, Tian M. Processing speed dysfunction is associated with functional corticostriatal circuit alterations in childhood epilepsy with centrotemporal spikes: a PET and fMRI study. Eur J Nucl Med Mol Imaging. 2022 Jul;49(9):3186-3196. doi: 10.1007/s00259-022-05740-w. Epub 2022 Feb 24. PMID 35199226